CLINICAL TRIAL: NCT04369846
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GM-XANTHO in Healthy Volunteers and to Investigate Its Efficacy and Safety Profile in Atopic Dermatitis Patients
Brief Title: A Phase I/IIa Study to Investigate the GM-XANTHO in Healthy Volunteers and Atopic Dermatitis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xantho Biotechnology Co., LTD (Industry)
Collaborators: Virginia Contract Research Organization Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: XANGMXA20160505
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test drug group (Experimental): The arm applies the test drug of GM-XANTHO
  Interventions: Drug: GM-XANTHO onitment
- Placebo group (Placebo Comparator): The arm applies the placebo
  Interventions: Drug: Placebo onitment

INTERVENTIONS:
Drug: GM-XANTHO onitment — Onitment application
  Other Names: Drawing blood
  Arms: Test drug group
Drug: Placebo onitment — Onitment application
  Other Names: Drawing blood
  Arms: Placebo group

SUMMARY:
A Phase I/IIa Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GM-XANTHO in Healthy Volunteers and to Investigate its Efficacy and Safety Profile in Atopic Dermatitis Patients

DETAILED DESCRIPTION:
The Phase I study is randomized, double-blind, placebo-controlled, dose escalating. There will be 3 dose cohorts, 4 (up to 8) subjects will be randomized in a 3:1 (GM-XANTHO to placebo) ratio in each cohort.The total study will take at least 23 days, conducted in National Taiwan University Hospital with 2-24 healthy subjects being enrolled.The Phase IIa study is randomized, double-blind, placebo-controlled, parallel. 2:1 ratio for GM-XANTHO to placebo control. The total study will take at least 43 days, conducted in National Taiwan University Hospital, Taipei Medical University Hospital, Ministry of Health and Welfare Shuang-Ho Hospital, and Linkou Chang-Gung Memorial Hospital with 102 Atopic Dermatitis patients being enrolled.

ELIGIBILITY:
Inclusion Criteria:

Phase I Number of patients achieving IGA of 0 or 1 with a ≥2 point improvement in Phase IIa study

* Female or male, age ≥ 20 years old
* Subjects whose body mass index (BMI) at screening is within a range of ≥ 18.5 kg/m2 and <30.0 kg/m2.

BMI = Body Weight (kg) / [Height (m) × Height (m)]2

* Subject's medical history shows no contraindication to the test medications.
* Subjects judged to be in good health by the investigator based upon the results of physical examinations (PEs), electrocardiogram (ECG) test, and all items of routine laboratory tests, including serum biochemistry, hematology and urinalysis, are within normal range as judged by the site. Assessment items of blood biochemistry include albumin, total protein, total bilirubin, ALP, SGOT, SGPT, BUN, serum creatinine. Assessment items of hematology tests include RBC count, WBC with differential counts, hemoglobin, hematocrit and platelet count. Assessment items of urinalysis include pH, color, appearance, gravity, erythrocyte, leukocyte, glucose, protein, ketones and nitrite.
* Female subjects show negative pregnancy test results and all male and female subjects with child-bearing potential (between puberty and 2 years after menopause) should use at least any one of the appropriate contraception methods as shown in inclusion criteria #12 of phase IIa prior to the first study dose.
* Subjects did not take any of the following medications in the specified durations:

  * Exposure of test sites to topical medications within 14 days prior to the application of IPs
  * Any systemically-absorbed medication (excluding vitamins, food supplements, and hormone contraceptives for birth control) within 14 days prior to the first dose of the study
  * Any enzyme inducer/inhibitor and/or known hepatic or renal clearance-altering agents within 30 days prior to the first dose of the study
* Subjects are willing to comply with protocol-stated requirements, instructions and restrictions, followed by understanding and signing the written informed consent form.

Phase IIa

* Female or male, age ≥ 20 years old
* Subjects who are diagnosed of atopic dermatitis based on the Hanifin and Rajka Criteria.
* Subjects who are with IGA score between mild (2) to moderate (3) and the Eczema Area and Severity Indices (EASI) are ≤ 20.
* Subjects who have body surface area of atopic dermatitis involvement ≥2%, ≤ 40% (≤20% if 10% GM-XANTHO would be used).
* Subjects who agree discontinuation of all treatment modalities, such as topical antihistamines, topical antimicrobials, topical corticosteroid and light treatments during the study treatment period for/on the affected site(s) (except the rescue medication prescribed by the study investigator(s)).
* Subjects who agree discontinuation of systemic corticosteroids, systemic antihistamines, and systemic immune-modulating agents during the study treatment period (except the standard medication oral antihistamine levocetirizine and rescue medication prescribed by the study investigator(s)).
* Subjects who are required to stop using treatment drugs listed in criteria# 5 for at least 14 days (or longer if the treatment half-life requires so; 7 half-lives should have elapsed) and treatment drugs listed in criteria# 6 for 28 days before the first investigational drug dose administration.
* Subjects who are judged to be in general good health (without clinically significant abnormalities) by the Investigator based on medical history, PEs, ECG, and routine laboratory tests at screening.
* Subjects who stopped immunosuppressant drugs for at least 28 days prior to the first dosing.
* Subjects who have taken oral antihistamine of levocetirizine 5mg once daily for at least 7 days before initiating the study treatment.
* Subjects who are eligible and able to participate in the study and accept to enter the study by signing this written informed consent form.
* If Subjects are male patients or female patients with child-bearing potential (between puberty and 2 years after menopause), subjects should use at least any one of the appropriate contraception methods shown below, for during and at least 4 weeks after GM-XANTHO treatment.

  1. Total abstinence (when this is in line with subjects preferred and usual lifestyle. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception).
  2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In the case of oophorectomy alone, subjects reproductive status should have been confirmed by follow up hormone level assessment.
  3. Male sterilization. Female patients' vasectomized male partner should be the sole partner.
  4. Combination of any two of the following listed methods: (d.1+d.2 or d.1+d.3, or d.2+d.3):

  d.1 Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example, hormone vaginal ring or transdermal hormone contraception.

  d.2 Placement of an intrauterine device (IUD) or intrauterine system (IUS). d.3 Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Exclusion Criteria:

Phase I:

* Subjects with the following conditions at the application site(s) that would interfere with the IP administration, skin assessment, or reaction to IPs:

  * presence of open sores
  * obvious differences in skin color between applications sites
  * excessive hair
  * scar tissue tattoo
  * coloration
* Subjects with any properly diagnosed disease within 30 days prior to the first dose of the study
* Subjects with any diagnosed dermatological or allergic diseases within 180 days prior to the first study dose
* Subjects with any clinically significant hematological, endocrine, cardiovascular, hepatic, renal, gastrointestinal, and/or pulmonary disorder; subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism and excretion of drugs
* Subjects had participated in investigational drug trials and took any investigational drug within 60 days prior to the first study dose.
* Subjects had blood donation for more than 250 mL within 60 days or 500 mL within 90 days prior to the first study dose.
* Subjects had a history of drug abuse or alcohol abuse according to the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) criteria.
* Subjects cannot stop smoking and caffeine-intakes for 48 hours prior to the first study dose and during the entire study period, and 48 hours after the last dose administration of IPs.
* Subjects who are inappropriate to participate in this study, as judged by the clinical Investigator
* Subjects who have been tested positive for the following tests:

  * Human immunodeficiency virus (HIV)
  * Hepatitis B virus (HBV): HBsAg and anti-HBc
  * Hepatitis C virus (HCV)

Phase IIa:

* Subjects who have participated in investigational drug trials and took any investigational drugs within 30 days or within 5 half-lives of the investigational drugs prior to the screening visit.
* Subjects who have any concurrent skin condition that will interfere with the assessment of treatment.
* Subjects who have an active infection on the atopic dermatitis site(s) at baseline.
* Subjects who are inevitable to engage in activities involving excessive or prolonged exposure to sunlight.
* Subjects who have known hypersensitivity to the study medication.
* Subjects who are with chronic condition(s) which either is not stable or not well controlled.
* Subjects who have positive results for HBV, HCV or HIV screens
* Subjects who are pregnant or breast feeding.
* Subjects who carry history of malignancy of any organ system (other than cervical carcinoma in situ or localized prostate cancer) within 5 years prior to study entry.
* Subjects who are not suitable to participate in the trial as judged by the Investigator(s).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
treatment emergent adverse events (TEAEs) | 7 days for Phase I
  Number of treatment emergent adverse events (TEAEs) occurring during the Phase I
IGA | 28 days for Phase IIa
  Number of patients achieving IGA of 0 or 1 with a ≥2 point improvement in Phase IIa study

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Ministry of Health and Welfare Shuang-Ho Hospital, New Taipei City, New Taipei
  - National Taiwan University Hospital, Taipei, Taipei
  - Taipei Medical University Hospital, Taipei, Taipei
  - Linkou Chang-Gung Memorial Hospital, Taoyuan District, Taoyuan

IPD SHARING:
Plan to Share IPD: No